CLINICAL TRIAL: NCT02057900
Title: Transplantation of Human Embryonic Stem Cell-derived CD15+ Isl-1+ Progenitors in Severe Heart Failure
Brief Title: Transplantation of Human Embryonic Stem Cell-derived Progenitors in Severe Heart Failure
Acronym: ESCORT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100303
Record Dates: First submitted 2013-09-17; First posted 2014-02-07 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Ischemic Heart Disease
Keywords: Postinfarction heart failure; Transplantation of human embryonic stem cell-derived cardiac progenitors; Tissue-engineered cellular graft; Fibrin hydrogel
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human embryonic stem cell (Experimental): Patients with ischemic heart failure receiving a fibrin gel embedding human embryonic stem cell-derived CD15+ Isl-1+ progenitors in addition to coronary artery bypass grafting and/or a mitral valve procedure.
  Interventions: Biological: Human embryonic stem cell-derived CD15+ Isl-1+ progenitors

INTERVENTIONS:
Biological: Human embryonic stem cell-derived CD15+ Isl-1+ progenitors — Epicardial delivery of a fibrin patch embedding human embryonic stem cell-derived CD15+ Isl-1+ progenitors

SUMMARY:
The purpose of the study is to assess the feasibility and safety of a transplantation of cardiac-committed progenitor cells derived from human embryonic stem cells in patients with severe heart failure.

DETAILED DESCRIPTION:
Heart failure due to coronary artery disease is a major problem because of its high prevalence, increased incidence and associated costs. When conventional medical/interventional treatments fail and if cardiac transplantation is contra-indicated, alternate options need to be considered. Transplantation of stem cells has emerged as one of them. While the optimal cell type still remains debatable, there is compelling evidence that cells whose phenotype closely matches that of the recipient tissue look sound candidates. In this context, human embryonic stem cells are attractive because of the possibility to drive their fate in vitro, prior to transplantation, towards a cardiac phenotype. We have developed a process for achieving such a commitment and generating cardiac-directed cells. The objective of this study is to assess both the feasibility and safety of this approach. In addition, the disadvantages of multiple intramyocardial injections have now been recognized. We have then taken advantage of the surgical setting of the trial (which entails concomitant coronary artery bypass or a mitral valve procedure) to switch from injections to the epicardial delivery of a fibrin gel into which the progenitor cells have been embedded. Coverage of this cell-loaded patch by an autologous pericardial flap is finally designed to provide trophic factors to the underlying cellular graft with the hope of improving its viability.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and less than 81 years
* Severe left ventricular systolic dysfunction with left ventricular ejection fraction (LVEF) ≤ 35% as assessed by echocardiography or scintigraphy
* History of myocardial infarction (older than 6 months) with a residual akinesia involving more than 2 (out of 16) contiguous segments, as assessed by basal echocardiography
* New York Heart Association (NYHA) Class III or IV despite optimal standard of care including diuretics and angiotensin receptor blockers and, if possible, beta blockers and aldosterone blockers
* Previous implantation of an automatic internal defibrillator associated, whenever indicated, to ventricular resynchronization
* Indication for a conventional cardiac surgical procedure : coronary artery bypass grafting involving, or not, the infarct area planned to be covered by the cell-loaded patch or mitral valve repair or replacement for ischemic mitral valve regurgitation; Non Eligibility to heart transplantation; Affiliation to a social security regimen
* Willingness and ability to give written informed consent

Exclusion Criteria:

* Pregnant or potentially child-bearing women
* Patients with poor echogenicity
* Left ventricular aneurysm
* Contra-indication to immunosuppressive drugs (history of cancer, infections like B or C hepatitis, positivity for Hepatitis-B, HIV, HTLV1)
* Contra-indication to sternotomy
* Alloimmunisation against the cell line from which the progenitors are derived
* Cardiogenic shock or NYHA Class IV heart failure requiring need for intravenous drugs
* Intellectual deterioration or psychiatric disease interfering with the ability to obtain an informed consent and to achieve a close follow-up of the patient
* Noncardiac disease which may reduce life expectancy in the short term
* Simultaneous participation to another trial

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05-27 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
number and nature of adverse events | Within the first year after surgery
  Evidence for new clinical/biological abnormalities, occurrence of arrhythmias or development of a cardiac or extra-cardiac tumor.

SECONDARY OUTCOMES:
Feasibility of patch's generation and its efficacy on cardiac functions | Within the first year after surgery
  Feasibility will be assessed by the ability to generate hESC-derived CD15+ Isl-1+ progenitors according to preset quality measures, to incorporate these cells in a fibrin patch, to deliver this patch onto the epicardium of the infarct area and to cover it with an autologous pericardial flap. Efficacy will be assessed on the following end points : 1- left ventricular function; 2- viability of the grafted area; 3- functional status; 4- major adverse cardiovascular events.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Menasché, MD, PhD, Principal Investigator — Department of Cardiovascular Surgery, Hôpital Européen Georges Pompidou, Paris, France
Locations (1):
- Department of Cardiovascular Surgery, Paris, France

REFERENCES:
- [Result] Puymirat E, Geha R, Tomescot A, Bellamy V, Larghero J, Trinquart L, Bruneval P, Desnos M, Hagege A, Puceat M, Menasche P. Can mesenchymal stem cells induce tolerance to cotransplanted human embryonic stem cells? Mol Ther. 2009 Jan;17(1):176-82. doi: 10.1038/mt.2008.208. Epub 2008 Oct 7. PMID 18841094
- [Derived] Menasche P, Vanneaux V, Hagege A, Bel A, Cholley B, Parouchev A, Cacciapuoti I, Al-Daccak R, Benhamouda N, Blons H, Agbulut O, Tosca L, Trouvin JH, Fabreguettes JR, Bellamy V, Charron D, Tartour E, Tachdjian G, Desnos M, Larghero J. Transplantation of Human Embryonic Stem Cell-Derived Cardiovascular Progenitors for Severe Ischemic Left Ventricular Dysfunction. J Am Coll Cardiol. 2018 Jan 30;71(4):429-438. doi: 10.1016/j.jacc.2017.11.047. PMID 29389360